CLINICAL TRIAL: NCT05150730
Title: "Self-perceived Health, Pain Intensity, and Work Ability of Individuals With Chronic Work-related Musculoskeletal Disease Followed up in a Multidisciplinary Care Program."
Brief Title: Individuals With Chronic Work-related Musculoskeletal Disease a Multidisciplinary Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Rosimeire Simprini Padula, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.135.916
Record Dates: First submitted 2021-11-21; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Musculoskeletal Diseases; Work-Related Condition; Chronic Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Chronic Pain

STUDY DESIGN:
Intervention Model Description: One group (n=88) of participants has analyzed pre and post-intervention. In total six groups with 10 to 19 participants each, participated in a multi-professional care program, held over the years 2017 and 2018. The care program had between 16 and 21 meetings, which took place once a week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality-of-Life multidisciplinary care program (Experimental): Six groups (between 10 -19 participants per group) received a meeting for two hours, the first hour being devoted to physical exercise, stimulating body awareness, improving mobility and muscle strengthening, relaxation and self-care.
  Interventions: Other: Multi professional care

INTERVENTIONS:
Other: Multi professional care — Participants were instructed to respect their pain threshold during body practice and the evolution of the participants happened gradually and individually. Associated with the practice of exercise, workers received information about their disease, chronic pain, guidelines for daily activities, and the importance of physical exercise. In the second hour, the responsible psychologist addressed issues such as the repercussions of illnesses on the individual's social and affective life, self-esteem, self-image, conformism, and self-indulgence after the illness and prospects for the future. Throughout the program, participants also received informative lectures from other professionals, such as social workers, nurses, and dentists.

SUMMARY:
Rehabilitation for work-related musculoskeletal disorders involves physical, behavioral, psychological treatment and counseling on how to deal with pain and disability. The study aims to evaluate the profile and indicators on the perception of health, pain intensity, and work ability (WA) of disability with work-related chronic musculoskeletal disease, assisted in a multidisciplinary program of worker health care.

DETAILED DESCRIPTION:
The study design is an intervention pre and post, 88 individuals diagnosed with work-related musculoskeletal disorders were followed up during a multidisciplinary program at the Reference Center for Workers' Health of the Unified Health System (SUS), SP, Brazil. The study was carried out six groups of individuals were followed (16 to 21 meetings; 10 to 19 participants). Sociodemographic, occupational, general health, pain intensity, and work ability (WA) were assessed at the baseline. Participants included has work-related musculoskeletal disorders diagnosis and complaints of chronic pain in one or more regions of the body, of different age groups, education levels, income, and occupational status (unemployed, leave work, or is working). Chronic pain is defined as a persistent or recurrent symptom lasting longer than three months. Criteria whose main diagnosis was a work-related mental disorder or musculoskeletal complaints related to previous injuries resulting from an accident or typical displacement from work, such as amputations and fractures, were excluded.

Outcome measure

1. Pain complains - Body region The diagnoses of musculoskeletal diseases were grouped by body segments: cervical spine, lumbar spine, upper limbs and lower limbs. Pain complaints reported by individuals were also grouped by segments: cervical, lumbar, more than one spinal segment, upper limbs, lower limbs, two areas of the body, three or more body region.
2. Pain intensity To measure pain intensity, the Numerical Rating Scale was used, an instrument that presents itself as a numbered line from zero (no pain) to ten points (maximum pain). Individuals responded about pain in the last seven days and in the last month.
3. Work ability - using two questions (current and future work ability). Based on the Work Ability Index (WA) have been inserted into this script questions about health perception, current and future WA (two years from now).
4. Emotional State
5. Job Satisfaction

   Two questions were also added to assess emotional state and job satisfaction. A Likert scale from 0 to 10 was used to answer all questions, and for the perception of health, current WA, future WA, and emotional state, the extremes represented respectively "very bad" and "great", and for satisfaction, 0 meant "totally dissatisfied" and 10 "totally satisfied".
6. Work demand The work demand was also evaluated based on the individual's perception of their work, in which they could refer to a greater physical or mental demand or the perception that their work involved both physical and mental demand, without any predominance.

ELIGIBILITY:
Inclusion Criteria:

* Participants included has work-related musculoskeletal disorders diagnosis and complaints of chronic pain in one or more regions of the body, of different age groups, education levels, income, and occupational status (unemployed, leave work, or is working). Chronic pain is defined as a persistent or recurrent symptom lasting longer than three months.

Exclusion Criteria:

* Participants whose main diagnosis was a work-related mental disorder or musculoskeletal complaints related to previous injuries resulting from an accident or typical displacement from work, such as amputations and fractures, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Frequency of Musculoskeletal complains | baseline, and through study completion, 1 year (12 months).
  Body region - The complaints reported by the individuals were also grouped by regions: cervical, lumbar spine, more than one segment of the spine, upper limbs, lower limbs, two body region, and three or more regions.
Values of Pain intensity | baseline, and at study completion, 1 year (12 months).
  Numeric Rating Scale - is a line numbered from zero (no pain) to ten points (maximum) pain). Individuals responded about pain in the last seven days and in the last month.
Values of Self-perceived Health | baseline, at study completion, 1 year (12 months).
  A Likert scale from 0 ("very bad") to 10 ("great")
Values of Work ability - current and future | baseline, and at study completion, 1 year (12 months).
  A Likert scale from 0 ("very bad") to 10 ("great")
Values of Emotional status | baseline, and at study completion, 1 year (12months).
  A Likert scale from 0 ("very bad") to 10 ("great")
Values of Job satisfaction | baseline, and at study completion, 1 year (12 months).
  A Likert scale from 0 totally unsatisfied" to 10 "totally satisfied".
Values of Pain intensity | baseline, and two months at the end of intervention (14 months) .
  Numeric Rating Scale - is a line numbered from zero (no pain) to ten points (maximum) pain). Individuals responded about pain in the last seven days and in the last month.
Values of Self-perceived Health | baseline, and two months at the end of intervention (14 months).
  A Likert scale from 0 ("very bad") to 10 ("great")
Values of Work ability - current and future | baseline, and two months at the end of intervention (14 months).
  A Likert scale from 0 ("very bad") to 10 ("great")
Values of Emotional status | baseline, and two months at the end of intervention (14 months).
  A Likert scale from 0 totally unsatisfied" to 10 "totally satisfied".
Values of Job satisfaction | baseline, and two months at the end of intervention (14 months).
  A Likert scale from 0 totally unsatisfied" to 10 "totally satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- Rosimeire Simprini Padula, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No